CLINICAL TRIAL: NCT05464641
Title: Total Knee Arthroplasty With Attune S+ or NexGen CR Randomised Study of 150 TKR
Brief Title: Randomised Total Knee Arthroplasty With Attune S+ or NexGen CR
Acronym: NexGe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Attune S+ or NexGen CR
Record Dates: First submitted 2022-03-24; First posted 2022-07-19 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: Knee arthroplasty

STUDY DESIGN:
Intervention Model Description: preoperative and 2 year postoperative
Who Masked: Participant
Masking Description: preoperative and 2 year postoperative
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- preoperative (Active Comparator): preoperative The Oxford Knee Score (OKS) is a 12-item patient-reported PRO, low score worse.
  Interventions: Other: Oxford knee score
- postoperative (Active Comparator): postoperative The Oxford Knee Score (OKS) is a 12-item patient-reported PRO, low score worse.
  Interventions: Other: Oxford knee score

INTERVENTIONS:
Other: Oxford knee score — The Oxford Knee Score (OKS) is a 12-item patient-reported PRO, low score worse

SUMMARY:
The primary purpose of this study is to evaluate the clinical performance of the Attune S+ knee primarily based on evaluation with use of Oxford Knee Score. The NexGen TKR will be used as reference standard. The second aim is to study component migration with model-based RSA in a subgroup of patients with model-based RSA and to compare these measurements with migration measurements with use of CT-based migration measurements. The investigators hypothesis is that the results two years after insertion of these two TKR designs will be about equal.

DETAILED DESCRIPTION:
The Attune knee was launched in 2012. From a clinical point of view some studies indicate superior clinical performance of the Attune when compared to the PFC. Carey and Harty operated 21 patients with both the Attune and the POFC Sigma knees. At six months' clinical scores were superior for the Attune side as was range of movement. Ranawat 2017, matched 100 Attune to 100 PFC Sigma knee operations based on age, gender, side and BMI but found no difference in clinical results after 2 years.

Bonutti reviewed three hospital databases and described 2 cases with loosening of the tibial component due to debonding between the cement and the implant, but the total material from which these cases were collected was not known or mentioned. Turgeon studied the fixation of 30 consecutive cases operated with the Attune knee and observed a mean maximum total point motion of 0.08 mm between 12 and 24 months, which suggests an acceptably low risk of medium to long-term failure due to aseptic loosening. Staats evaluated incidence of radiolucent lines in 276 Attune and 253 PFC Sigma TKRs up to one year after operation and observed a higher incidence in the former group.

In the last report from NJR from 2020, the 5-year revision rate of the Attune FB knee is 2.71 (2.32-3.17), which is slightly above average (2.23, 2.20-2.26). In the Australian registry from 2020 the corresponding cumulative percent revision rate of cemented Attune CR is 3.0 % (2.7 - 3.5) at 5 years.

In an ongoing study the investigators have randomized 95 knees with knee osteoarthritis to either become operated with an Attune knee (n=49) or a PFC knee (n=46). Preliminary results at one year show almost equal results when evaluated in terms of Oxford Knee or Forgotten Joint Scores.

NexGen metal-backed tibia is the most commonly used total knee prosthesis in Sweden. Its revision rate is one of the lowest observed in the Swedish Register. The 5 years survival in the report from NJR from 2020 is 2.1% (2.05 - 2.21) and in the report from the Australian register it is about equal (2.0; 1.9 - 2.2). The Australian Register also present survival at 19 years amounting to 5.7% (4.7 - 6.9) being the lowest cumulative revision of those specific cemented TKRs accounted for with that long follow up.

In 2017 DePuy launched the Attune S+ tibial components in order to address the potential problem of loosening between the cement and the tibial tray. If and if so, to what extent this modification will change the clinical outcome of TKRs operated with this implant is not known. Based on the high survival rate of the in Sweden frequently used NexGen TKR a comparative study between the Attune S+ and the NexGen TKRs would provide an important benchmark for the performance of the Attune S+ knee.

ELIGIBILITY:
Inclusion Criteria:

* Medial or lateral primary OA Ahlbäck Grade 2-4
* Varus or valgus deformity ≤10 degrees, extension defect ≤10 degrees
* Age 40-75 years
* BMI <35
* ASA 1-3.
* Coming from independent living in own home
* Written informed consent.

Exclusion Criteria:

* Cortisone treatment during the last 6 months before operation
* Neurological diseases with symptoms, stroke with sequel
* Endocrine diseases with symptoms
* OA secondary to trauma, infection, inflammatory disease or congenital and acquired deformities
* BMI >=35

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Oxford knee score | preoperative
  Oxford knee score, a 12-item patient-reported PRO
Oxford knee score | 2 year postoperative
  Oxford knee score, a 12-item patient-reported PRO

CONTACTS AND LOCATIONS:
Overall Officials: Roland Zügner, PhD, Principal Investigator — Göteborg University
Locations (1):
- Roland Zügner, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No
upon request